CLINICAL TRIAL: NCT02060643
Title: A Cross-sectional Study Looking at the Effect of Radiotherapy on Carotid Intima-medial Thickness in Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Royal Brompton and Harefield NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCR 3687
Record Dates: First submitted 2014-02-06; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Head and Neck Tumours

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cross-sectional hemi-neck RT

SUMMARY:
Some patients with head and neck cancer or benign tumours of the head and neck receive radiotherapy to their neck as part of their treatment. The carotid arteries are often included in the radiotherapy as collateral structures. There is some evidence to show that radiotherapy to these blood vessels can result in thickening of the artery walls some years after treatment and increased risk of stroke or TIA in the future.

Current research is now aimed towards detecting radiotherapy-related changes to the carotid arteries at an earlier stage and towards using new radiotherapy techniques to avoid treating these blood vessels if possible. The question of whether or not the use of preventive medicines like aspirin and cholesterol-lowering tablets helps to reverse this process is currently unanswered.

The aim of this study is to measure the thickness (intima-medial thickness) of irradiated carotid artery walls and compare this to unirradiated arteries. There are many other causes for thickening of arteries (such as high blood pressure, high cholesterol levels and diabetes) and these may affect the ability to measure the effect of radiotherapy change to the artery wall. In order to address this, it is ideal to look at this process in patients who have only had one side of their neck treated and use the other side as a comparison. The study will also be looking for earlier signs of radiotherapy-related changes, such as stiffening of the artery wall, inflammation in the artery wall (a very early sign of radiotherapy-related change) and some markers in the blood that may indicate that this process is taking place.

The null hypotheses of this study are:

* In irradiated carotid arteries, the mean intimal-medial thickness will be the same compared to unirradiated arteries.
* Serum biomarkers will not be elevated in radiation-induced carotid atherosclerosis.
* Development of radiation-induced carotid atherosclerosis is not affected by risk factor modulation (Aspirin, HMGCoA reductase inhibitors, smoking cessation).
* There is no difference in carotid arterial wall strain in irradiated carotid arteries versus unirradiated carotid arteries.
* Microbubble ultrasound will not be able to detect Inflammation in the carotid arteries as an early marker of atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Histologically confirmed cancer or benign tumours of the head and neck area treated with hemi-neck radiotherapy to ≥ 50Gy
* Received radiotherapy to the neck area more than 24 months previously
* Intervening neck dissection allowed
* Be able to provide written informed consent

Exclusion Criteria:

* Patients who have active head and neck cancer
* Patients with a prior history of carotid endarterectomy or carotid angioplasty and stenting

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with histologically confirmed cancer or benign tumours of the head and neck area treated with hemi-neck radiotherapy to ≥ 50Gy
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The difference in mean IMT between irradiated and unirradiated carotid arteries. | >2 years post-radiotherapy
  Cross-sectional study - measured at one time-point at least 2 years after radiotherapy

SECONDARY OUTCOMES:
The prevalence of carotid artery stenosis in irradiated carotid arteries compared to unirradiated carotid arteries. | >2 years post-radiotherapy
  Cross-sectional - measured at one time point at least 2 years after radiotherapy
Quantify the use of risk-modifying therapy (anti-hypertensives, anti-diabetic medication, HMGCoA reductase inhibitors, smoking cessation) and their effect on radiation-induced carotid atherosclerosis. | > 2 years post-radiotherapy
  Cross-sectional - measured at one time point at least 2 years after radiotherapy
Correlation of serum biomarker levels to carotid IMT and strain. | > 2 years post-radiotherapy
  Cross-sectional - measured at one time point at least 2 years after radiotherapy
The difference in arterial wall strain between irradiated and unirradiated carotid arteries | > 2 years post-radiotherapy
  Cross-sectional - measured at least 2 years after radiotherapy
The difference in arterial wall inflammation between irradiated and unirradiated carotid arteries | > 2 years post-radiotherapy
  Cross-sectional - measured at one time point at least 2 years after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Nutting, PhD, Principal Investigator — Royal Marsden NHS Foundation Trust